CLINICAL TRIAL: NCT04468555
Title: Effects of Global Postural Reeducation on Hallux Valgus
Brief Title: Hallux Valgus Manual Therapy Based on Global Postural Reeducation.
Acronym: HVMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, DAVID CRUZ DÍAZ, Professor, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HVUJA
Record Dates: First submitted 2020-07-04; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Hallux Valgus; Hallux Deformity; Foot Deformities
MeSH Terms: conditions — Hallux Valgus; Foot Deformities

STUDY DESIGN:
Intervention Model Description: A single-blind randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent assessor blinded to the data collection was responsible for the allocation process. A list of the computer-generated number was employed to assign participants to experimental or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Global postural reeducation (Experimental): Patients completed 3 sessions of global postural reeducation for 3 weeks.
  Interventions: Other: Global postural reeducation
- Control group (No Intervention): Patients allocated to the control group did not receive any treatment.

INTERVENTIONS:
Other: Global postural reeducation — It consisted of Global Postural Re-Education sessions divided into 3 sessions and performed with a frequency of 1 per week for 3 weeks. The sessions were performed individually, with an approximate duration of 40 minutes and all of them were assessed by the same physiotherapist.
  Arms: Global postural reeducation

SUMMARY:
Manual approach of Hallux Valgus with global postural reeducation.

DETAILED DESCRIPTION:
Hallux Abducto Valgus is a frequent pathology with a prevalence of 30% in women and 13% in men. The tendency is to increase with age.

Usually, the elected treatment is surgery, as the conservative orthopedic methods are used at the early stages of the pathology. Global Postural Re-Education is a manual therapy treatment method through which we can treat lots of pathologies. Some investigations demonstrate Postural Re-Education is effective for the treatment of temporomandibular disorders, urinary incontinence, and spine disorders, but there is no scientific evidence that defends the improvement of the symptoms and correction of the angle of the Hallux Abducto Valgus using Postural Re-Education.

ELIGIBILITY:
Inclusion Criteria:

* hallux abducto valgus with an angle between 15 - 39º
* pain on the medial or plantar face of the forefoot
* Physical independence to take part in the study.

Exclusion Criteria:

* Being under hallux abducto valgus treatment.
* Lower limb surgery.
* Fracture or disfunction on the lower limb other than hallux valgus which may affect the studied variables.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Postural control | From baseline to 3 weeks and 8 weeks.
  Postural control was evaluated by means of a stabilometric platform of resistive pressure sensors (Sensor Medica, Rome, Italy). There will be performed two tests: open eyes Romberg and closed eyes Romberg.

SECONDARY OUTCOMES:
Dynamic balance | From baseline to 3 weeks and 8 weeks.
  Dynamic balance has been measured by a simplified version of the Star Excursion Balance Test where the anterior, posteromedial and posterolateral reach directions were collected for statistical analysis.
Ankle range of motion | From baseline to 3 weeks and 8 weeks.
  Ankle dorsiflexion range of motion was assessed by the weight-bearing lunge test. The patient is positioned in a standing position facing a wall with the involved foot parallel with a tape measure which has been attached to the floor and the opposite leg placed behind in a tandem stance. A forward lunge is performed until the anterior knee tries to make contact with the wall with the heel firmly planted on the ground.
Self-reported instability | From baseline to 3 weeks and 8 weeks.
  To determine the severity of ankle instability the Cumberland ankle instability tool was used. The total score of the nine items ranges from 0 (severe instability) to 30 (normal stability).
Assessment of the grade of hallux valgus | From baseline to 3 weeks and 8 weeks.
  With the Manchester Scale the examiners grade the feet of the participants in: A: no hallux valgus; B: mild hallux valgus; C: moderate hallux valgus; D: severe hallux valgus.
Foot posture | From baseline to 3 weeks and 8 weeks.
  it will be performed the Foot Posture Index 6-items for evaluating the general foot position. It is graded as pronated, neutral or supinated depending on the punctuation
Passive and active dorsiflexion range of motion of the 1st metatarsophalangeal joint | From baseline to 3 weeks and 8 weeks.
  it will be assessed by the Jack test, in which the phalangeal bone is passively dorsiflexed and the plantar arch is observed. The aim is classified the Windlass Mechanism in: intact; limited; absent. The active range of motion will be assessed by kinovea software.
Gait parameters | From baseline to 3 weeks and 8 weeks.
  Gait parameters after treatment with optogait system including gait cycle, contact time, flight time, and pre-swing phase during walking and running.
Functional status | From baseline to 3 weeks and 8 weeks.
  Function in daily living and sport activities were assessed by the Foot and Ankle Ability Measure. This questionnaire Is divided by two subscales of 21 items (daily living subscale) and 8 items (sports subscale). The obtained score is expressed as a percentage calculated by dividing the patient's score by max score and the lower percentage is related to the lower level of function.

CONTACTS AND LOCATIONS:
Overall Officials: David Cruz-Diaz, PhD, Study Director — University of Jaén
Locations (1):
- University of Jaen, Jaén, Spain